CLINICAL TRIAL: NCT07172945
Title: Research and Follow-up of the Determinants of the Progression and Complications of Inflammatory Bowel Diseases Treated or Not With Immunosuppressants
Acronym: SUIVITHEQUE2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Sorbonne University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP240151; IDRCB: 2024-A00348-39 (Other: ANSM)
Record Dates: First submitted 2024-11-21; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Crohn; Ulcerative Colitis (UC); IBD (Inflammatory Bowel Disease)
Keywords: Microbiome; Biobank; Crohn; Ulcerative colitis; IBD
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Blood Specimen Collection; Defecation; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients with Inflammatory Bowel Diseases (Other)
  Interventions: Other: Blood, fecal, saliva; Other: intestinal content samples and biopsies
- Microbiota control' subjects (Other)
  Interventions: Other: Blood, fecal, saliva
- Endoscopy control' subjects (Other)
  Interventions: Other: Blood, fecal, saliva; Other: intestinal content samples and biopsies

INTERVENTIONS:
Other: Blood, fecal, saliva — Blood, fecal and saliva samples
Other: intestinal content samples and biopsies — intestinal content samples and biopsies obtained per upper or lower gastrointestinal tract endoscopy
  Arms: Endoscopy control' subjects; Patients with Inflammatory Bowel Diseases

SUMMARY:
Inflammatory Bowel Diseases (IBD), including Crohn's disease (CD) and ulcerative colitis (UC), are chronic, disabling conditions affecting young adults, marked by flare-ups and remissions. Traditionally, IBD was treated with immunosuppressants like thiopurines, but new biological treatments, such as anti-TNFa antibodies (e.g., infliximab, adalimumab), have transformed management. Biologics often combine with thiopurines but come with risks, like increased chances of skin cancers and lymphomas, especially for prolonged use in young patients. Recently, newer biologics (e.g., ustekinumab, vedolizumab) and small molecules like JAK inhibitors have expanded treatment options.

The exact cause of IBD remains unknown, though an inappropriate immune response to the intestinal microbiota in genetically predisposed individuals is suspected. Dysbiosis, or imbalance in gut microbiota, has been linked to IBD, with reductions in 'beneficial' bacteria and increases in harmful ones. Certain bacteria, like Faecalibacterium prausnitzii, may serve as markers for disease activity or progression.

Due to the heterogeneity of UC and CD, it is crucial to identify early predictive factors for complications and treatment response. This study aims to identify biological markers of disease course and complications in IBD and to deepen understanding of its pathophysiological mechanisms.

DETAILED DESCRIPTION:
Inflammatory Bowel Diseases (IBD) are chronic, disabling conditions that affect young adults with a predilection for flare-ups interspersed with periods of remission. Crohn's disease (CD) and ulcerative colitis (UC) are the two main types of IBD.

IBD is a chronic disease, the course of which is often marked by complications. Until recently, the medical treatment of IBD was based on the use of immunosuppressants, particularly thiopurines. The management of IBD has been modified in recent years by the appearance of new so-called 'biological' treatments. Anti-TNFa antibodies (such as infliximab or adalimumab) represent, highly effective weapon in the arsenal available for treating IBD. Biological treatments appear to have a synergistic effect with thiopurines and their administration is therefore often concomitant. These immunosuppressive and biological treatments are not harmless, especially as they are taken for prolonged periods by young patients. In particular, the use of thiopurines is associated with a marked increase in the risk of non-melanoma skin cancers and lymphomas. The long-term risks of biological treatments are still poorly understood. For the treatment of IBD, there are now much more biologics available, including Ustekinumab, vedolizumab and also small molecules, such as JAK inhibitors.

Despite recent advances, the cause of IBD remains unknown. The currently dominant hypothesis is that of an inappropriate immune response to the intestinal microbiota in genetically predisposed individuals.

In humans, an imbalance in the composition of the intestinal microbiota (dysbiosis) has been demonstrated in patients with CD and UC, with a reduction in 'beneficial' bacteria and an increase in potentially 'harmful' bacteria. Finally, certain bacteria in the intestinal microbiota could be used as a marker of disease activity or as a predictive factor for progression, as we have shown with the Faecalibacterium prausnitzii bacterium and postoperative recurrence of Crohn's disease.

Given the phenotypic heterogeneity of UC and CD in terms of progression and complications, it is essential to identify predictive factors that will enable patients at risk to be identified as early as possible so that treatment can be adapted at an early stage.

Given the clinical and pathophysiological heterogeneity of IBD, it would seem difficult to use clinical factors alone to predict patient outcome. On the other hand, it would also be very important to be able to predict the response or side-effects of a treatment before starting it, which again would enable appropriate decisions to be made without wasting time. It therefore seems necessary to look for biological determinants of the course and complications of IBD.

The aims of the study are (i) to identify biological determinants of the course, complications and response to treatment of chronic inflammatory bowel disease and (ii) to gain a better understanding of the underlying pathophysiological mechanisms.

The primary outcome is to describe the Biological parameters of the host and microbiota as a prognosis factor, and the response to treatment in IBD.

The secondary outcomes are lister below:

* Identification of genetic polymorphisms
* Identification of serum markers
* Identification of iImmune characteristics of the intestinal microbiota
* Identification of markers of the intestinal microbiota
* Mucosal characteristics of the intestinal microbiota
* Mucosal markers of the intestinal microbiota
* Mechanistic analysis: Exploratory study into the pathophysiology of host-microbiota interactions; interactions between epithelial cells, immune cells and micro-organisms and omics analysis including microbiome sequencing, transcriptomics, metabolomics, and functional assay will be perform to analyze the interactions between epithelial or immune cells with the gut microbiome

ELIGIBILITY:
Inclusion Criteria:

For all patients and control subjects

* Person able to give free and informed consent.
* Age ≥ 18 years.
* Beneficiary of a social protection scheme or entitled person (excluding AME).
* Consultation in the Gastroenterology and Nutrition Department of Saint-Antoine Hospital

Patients with IBD :

- Patients with Crohn's disease or haemorrhagic rectocolitis with a diagnosis established or confirmed in the Gastroenterology and Nutrition Department at Saint-Antoine Hospital.

Microbiota control' subjects:

- Healthy subjects seen in consultation as a preventive measure or as part of stool donations for FMT.

Endoscopy control' subjects:

- Subjects with a medical indication for digestive endoscopy with biopsies:

* For upper endoscopy: moderate upper digestive symptoms such as epigastralgia or pyrosis
* For colonoscopy: moderate digestive symptoms suggestive of irritable bowel syndrome or screening for colorectal cancer.

Exclusion Criteria:

For all patients and control subjects

* Subjects under guardianship, curatorship or safeguard of justice.
* Subjects who do not speak French.

IBD patients:

- Colon preparation within 6 weeks before stool sampling (stool samples may be taken either before colonoscopy or at least 6 weeks afterwards).

Endoscopy control' and "microbiota control" subjects:

* Subject suffering from a chronic disease
* Antibiotics taken in the 6 weeks prior to endoscopy
* Antibiotics or colonic preparation taken within 6 weeks prior to stool sampling (stool samples may be taken either before colonoscopy or at least 6 weeks afterwards).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2040-11 (Estimated); Study Completion 2040-11 (Estimated)

PRIMARY OUTCOMES:
Relation between biological parameters (fecal and ileal microbiome) and outcomes of IBD | up to 12 months after the inclusion
  identify relations between fecal and ileal microbiome and disease evolution

CONTACTS AND LOCATIONS:
Overall Officials: Harry SOKOL, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Yes
plans to share these data outside the primary research group for secondary research purposes like re-analysis, secondary analysis, or meta-analysis. Data may be shared via an online platform, an email request, nonelectronic transfer, or other method